CLINICAL TRIAL: NCT07175155
Title: Combination of COMBO Endoscopy Oropharyngeal Airway and High-flow Nasal Cannula Oxygenation in Sedated Gastrointestinal Endoscopy for Morbidly Obese Patients: a Multicenter, Randomized, Controlled Clinical Trial
Brief Title: Combination of COMBO Endoscopy Oropharyngeal Airway and HFNC Oxygenation in Sedated Gastrointestinal Endoscopy for Morbidly Obese Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Diansan Su, Chief Physician,Researcher, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZJU2025C140
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-10

CONDITIONS: Hypoxemia; Esophageal Cancer; Morbidly Obese Patients; Gastric Cancer
Keywords: COMBO Endoscopy Oropharyngeal Airway; Hypoxemia; Sedation; Gastrointestinal Endoscopy; high-flow nasal cannula
MeSH Terms: conditions — Hypoxia; Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COMBO Endoscopy Oropharyngeal Airway with High-Flow Nasal Cannula Oxygenation (Experimental): In this group, patients use the COMBO Endoscopy Oropharyngeal Airway with High-Flow Nasal Cannula Oxygenation
  Interventions: Device: COMBO Endoscopy Oropharyngeal Airway with High-Flow Nasal Cannula Oxygenation
- High-Flow Nasal Cannula Oxygenation (Active Comparator): In this group, patients use the High-Flow Nasal Cannula Oxygenation
  Interventions: Device: High-Flow Nasal Cannula Oxygenation

INTERVENTIONS:
Device: COMBO Endoscopy Oropharyngeal Airway with High-Flow Nasal Cannula Oxygenation — Using the COMBO endoscopy oropharyngeal airway with High-Flow Nasal Cannula Oxygenation in sedated gastrointestinal endoscopy for morbidly obese patients
  Arms: COMBO Endoscopy Oropharyngeal Airway with High-Flow Nasal Cannula Oxygenation
Device: High-Flow Nasal Cannula Oxygenation — In this group, patients use high-flow nasal cannula oxygenation
  Arms: High-Flow Nasal Cannula Oxygenation

SUMMARY:
Hypoxaemia during sedated gastrointestinal endoscopy exceeds 40 % in morbidly obese (BMI ≥ 35 kg m-²) patients. High-flow nasal cannula alone often fails because of persistent airway collapse. A recent innovation in this domain is the COMBO Endoscopy Oropharyngeal Airway-a multifaceted device that encompasses capnography monitoring, bite block , oxygenation support, and oropharyngeal airway management.The purpose of this study is to investigate whether the combination of the COMBO Endoscopy Oropharyngeal Airway and High-Flow Nasal Cannula oxygenation reduces the incidence of hypoxemia in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* BMI ≥ 35 kg/m².
* Patients undergoing gastroscopy or gastrointestinal endoscopy.
* The estimated duration of the procedure does not exceed 45 minutes.
* Patients have signed the informed consent form.

Exclusion Criteria:

* Coagulation disorders or bleeding tendency (e.g., oral/nasal bleeding risk, mucosal injury, oropharyngeal obstruction) making oropharyngeal airway placement unsafe or unfeasible.
* Active upper respiratory tract infection (oral, nasal, or pharyngeal), or fever (core temperature >37.5°C).
* Chronic obstructive pulmonary disease or other acute/chronic pulmonary diseases requiring long-term or intermittent oxygen therapy, or preoperative SpO₂ ≤ 92% on room air.
* Severe organ dysfunction, including: Cardiac insufficiency (<4 METs), Severe renal insufficiency (requiring dialysis), Diagnosed severe hepatic insufficiency, Increased intracranial pressure, ASA physical status ≥ IV.
* Confirmed pregnancy or current breastfeeding.
* Known allergy to sedatives (e.g., propofol) or medical adhesives.
* Multiple traumatic injuries.
* Current participation in another clinical trial.
* Other conditions deemed unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2027-08-20 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxemia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  75% ≤ SpO2 < 90% for <60 s

SECONDARY OUTCOMES:
The incidence of sub-clinical respiratory depression | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  90% ≤ SpO2 < 95%
The incidence of severe hypoxaemia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  SpO2 < 75% or 75% ≤ SpO2 < 90% for ≥60 s

OTHER OUTCOMES:
The incidence of other adverse events | Patients will be followed for the duration of hospital stay, an expected average about 2 hours.
  Other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Jinjiang Municipal Hospital, Jinjiang, Fujian
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Fifth Affiliated Hospital of Wenzhou Medical University, Lishui, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided